CLINICAL TRIAL: NCT05434949
Title: Effect of Post-prandial State, Statins and PCSK9 Inhibitors on Serum 7a-hydroxy-4-cholesten-3-one Concentration
Brief Title: Pre-analytical Influences on a Blood Test Study
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022LAB126
Record Dates: First submitted 2022-06-01; First posted 2022-06-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Effect of food intake on C4: Blood tests to analyse serum C4 pre, and 2 and 4 hours post a standardised meal, and the same 10 patients to analyse serum C4 at 0, 2 and 4 hours, all fasting.
  Interventions: Diagnostic Test: Blood test
- Effect of Lipid-lowering therapy on C4: Spare sample collected from patients before and after starting on lipid-lowering therapy will be used to measure C4 before and after lipid-lowering therapy.
  Interventions: Other: Analyses of samples

INTERVENTIONS:
Diagnostic Test: Blood test — Three blood samples to be taken at 08.00, 10.00 and 12.00 on day 1 of the study.
  The following day, after an overnight fast, a blood sample will be taken at 8.00, followed by a standardized breakfast provided by the study team at 8.30, and then two further blood samples at 10.00 and 12.00.
  Groups: Effect of food intake on C4
Other: Analyses of samples — C4 will be measured in surplus serum from 30 adult lipid patients before starting on lipid-lowering therapy (either statin of PCSK9 therapy) and then again 3 months after starting on therapy. Blood samples will be collected as part of routine lipid management, no additional samples are required.
  Groups: Effect of Lipid-lowering therapy on C4

SUMMARY:
Chronic diarrhoea is common and often believed to result from irritable bowel syndrome (IBS). However, up to 50% of patients with an IBS diagnosis may have something called Bile Acid Diarrhoea (BAD) instead. BAD is easily treatable however diagnosis currently relies on a complex test involving two full body scans. The aim of the study is therefore to investigate whether a simple laboratory test, that can be done on a single blood sample, would be appropriate instead. This laboratory test is called 7aC4.

In order to determine whether 7aC4 could be a good test for BAD, it needs to be determined whether eating a meal can alter the levels of 7aC4. The aim of this study is to measure 7aC4 at several time points before and after eating a meal, to see what effect this has on 7aC4 levels.

DETAILED DESCRIPTION:
Chronic diarrhoea is common and largely due to irritable bowel syndrome (IBS). IBS is reported to affect about 11% of the UK population. About half these patients are believed, however, to have bile acid diarrhoea (BAD). There are, therefore, more than one million patients with BAD in the UK. BAD is caused by small bowel malabsorption of bile acids (BA) and increased BA in the large intestine cause diarrhoea. Once diagnosed, the treatment of BAD is simple and effective. BAD, however, is often not diagnosed because of a lack of easily available and reliable diagnostic methods.

In the UK, the radiolabelled 23-seleno-25-homotaurocholic acid test (SeHCAT) is the gold-standard diagnostic method. The SeHCAT is performed by oral administration of a radiolabel, followed by two full-body scans, one week apart, to assess retention of BA. A low retention time indicates BAD. SeHCAT, however, is expensive, inconvenient to the patient, exposes the patient to radiation and has limited availability. A simple laboratory biomarker for the diagnosis of BAD is, therefore, desirable.

Proposed diagnostic laboratory biomarkers for BAD include measurement of faecal BA and serum 7a-hydroxy-4-cholesten-3-one (C4). C4, an intermediate in the BA synthesis pathway, is the common precursor for the primary BAs. It is, therefore, utilised as a biomarker of BA synthesis. Serum C4 increases in BAD, as BA synthesis increases to compensate for the increased faecal BA loss. C4 measurement requires a single serum sample for analysis by liquid chromatography tandem mass spectrometry (LC-MS/MS). There is, however, limited data comparing its diagnostic accuracy to the SeHCAT scan. Furthermore, pre-analytical variables which may affect C4, include cholesterol lowering medication, diurnal variation and effects of food intake require clarification to optimise conditions for sample collection before its introduction into routine laboratory use. Literature suggests both diurnal variation and post-prandial response can influence C4 levels, however there is limited information on whether this is primarily a post-prandial response, or due to diurnal variation. This study aims to compare pre- and post-prandial C4 levels, controlled for diurnal variation.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Effect of food intake on C4

• Healthy adult (>=18 years) volunteers from the BCPS.

Part 2: Effect of Lipid-lowering therapy on C4

• There is no patient recruitment. Spare sample collected from patients before and after starting on lipid-lowering therapy will be used.

Exclusion Criteria:

Part 1: Effect of food intake on serum C4

* Subjects with learning disability or those lacking mental capacity to give consent.
* Pregnant or breast-feeding
* On (prescribed and over-the-counter) medication and herbal remedies known or considered to affect lipid and bile acid metabolism.
* Chronic and acute diarrhoea
* Gastrointestinal disease.
* Previous ileal resection or cholecystectomy
* Obesity defined as a body mass index (BMI) of greater than 29.9 kg/m2

Part 2: Effect of Lipid-lowering therapy on C4

The surplus serum will not be analysed if any of the following apply to the patient:

* Pregnant or breastfeeding for either time point
* Lipid lowering therapy within the last 6 months for the first sample
* On (prescribed and over-the-counter) medication and herbal remedies known or considered to affect lipid and bile acid metabolism.
* Chronic and acute diarrhoea
* Gastrointestinal disease.
* Previous ileal resection or cholecystectomy
* Obesity defined as a body mass index (BMI) of greater than 29.9 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers from the BCPS and patients attending hospital as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Serum C4 will be measured by liquid chromatography tandem mass spectrometry (LC-MS/MS) to measure increase/ decrease by diurnal variation and food intake. | 12 months
  Serum C4 will be measured by liquid chromatography tandem mass spectrometry (LC-MS/MS) to measure increase/ decrease by diurnal variation and food intake.
Measure increase/decrease in Serum C4 levels after taking lipid lowering therapy (statins / PCSK9 inhibitors). | 12 months
  Measure increase/decrease in Serum C4 levels after taking lipid lowering therapy (statins / PCSK9 inhibitors).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided